CLINICAL TRIAL: NCT02844673
Title: Effect of Mobile-Directly Observed Therapy (DOT) on Adherence to Hydroxyurea Treatment in Adult HbSS Patients at Muhimbili National Hospital (MNH) in Tanzania: a Pilot Study
Brief Title: Mobile-Directly Observed Therapy on Adherence to Hydroxyurea
Acronym: mDOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Collaborators: University of Pittsburgh (Other); Muhimbili National Hospital (Unknown)
Responsible Party: Principal Investigator, Ábel Makubi, Senior Lecturer, Muhimbili University of Health and Allied Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUPI-001
Record Dates: First submitted 2016-07-18; First posted 2016-07-26 (Estimated); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Anaemia
Keywords: Sickle cell disease; Hydroxyurea; Adherence; randomized trial; medication possession ratio
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard monitoring (SM) arm (Active Comparator): Participants will receive fixed dose hydroxyurea therapy (15 mg/Kg/day) with standard monitoring. Standard monitoring is defined as a follow-up visit two weeks after initiation of therapy and monthly follow-ups thereafter
  Interventions: Drug: Hydroxyurea
- mDOT arm (Experimental): Participants will receive fixed dose hydroxyurea therapy (15 mg/Kg/day) and Mobile Directly Observed Therapy (mDOT) consisting of a web based medication adherence monitoring system that includes direct video confirmation of adherence using the patient's personal cellular telephone. Participants will receive alerts on their cell phone at pre-arranged times to remind them to take their medications. Participants will be followed-up at two weeks after initiation of therapy and monthly thereafter.
  Interventions: Drug: Hydroxyurea; Device: Mobile Directly Observed Therapy

INTERVENTIONS:
Drug: Hydroxyurea — Patients will receive fixed dose Hydroxyurea therapy (15 mg/Kg/day) with standard monitoring
Device: Mobile Directly Observed Therapy — Mobile DOT will consist of a web based medication adherence monitoring system that includes direct video confirmation of adherence using the patient's personal cellular telephone. Patients will receive alerts on their cell phone at pre-arranged times to remind them to take their medications.
  Other Names: mDOT
  Arms: mDOT arm

SUMMARY:
To examine the effect of mobile-directly observed therapy (mDOT) on adherence to HU (mDOT-HuA) adults with SCA at Muhimbili National Hospital (MNH) in Tanzania.

DETAILED DESCRIPTION:
Background: Hydroxyurea (HU) has been demonstrated to be efficacious in reducing complications in individuals with Sickle Cell Anemia (SCA) but poor adherence is a barrier to improving outcomes in patients with SCA. Directly Observed Therapy (DOT) has been shown to improve adherence in various chronic diseases but there is limited data in adults with sickle cell anaemia (SCA).

Methods and design: To examine the effect of mobile-directly observed therapy (mDOT) on adherence to HU (mDOT-HuA) adults with SCA at Muhimbili National Hospital (MNH) in Tanzania.The mDOT-HuA study is single centre, prospective, randomized, open label clinical trial. 100 participants with SCA with hemoglobin SS genotype, aged ≥18 years, living in urban Dar es Salaam and able and willing to participate in the study. Participants will be divided into two treatment arms; 50 in standard monitoring (SM) arm: will receive fixed dose HU therapy with standard monitoring. 50 in treatment mDOT arm: will receive fixed dose HU therapy with standard monitoring and a mobile direct observed web based medication adherence monitoring system. The primary outcome is adherence to HU as defined as medication possession ratio of ≥80 at end of 3 months of HU treatment and mDOT monitoring. Secondary outcomes will be efficacy to HU treatment as measured through the the mean change in fetal hemoglobin (between baseline and end of 3 months) and safety, measured as the proportion of participants experiencing serious adverse events related to HU at week 2, 6, 10 and at the end of 3 months.

REDCap, an open source software application will be used to collect data using clinical research forms.

Conclusion: This project has the potential for the development of novel strategies for improving HU adherence in SCA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and living in urban Dar es Salaam
* Male or female (post-menopausal, sterile, or using an acceptable method of contraception)
* Negative urine pregnancy test at Screening and a negative urine pregnancy test (dipstick) prior to randomization and dosing
* Hemoglobin SS genotype
* Absolute neutrophil count >1,500/uL
* Platelet count >95,000/uL
* Serum creatinine< 100 µmol/L (1.2 mg/dL)
* Alanine transaminase (ALT) less than two times the upper limit of normal
* Being able and willing to record and submit videos electronically

Exclusion Criteria:

* Chronic transfusion program as defined by participating in a scheduled (pre-planned) series of transfusions for prophylactic purposes or has a hemoglobin A level that is >20% of the total hemoglobin
* Hemoglobin <4.0 g/dL
* HIV positive
* Female planning to become pregnant during the study period
* Serious mental (including psychosis) or physical illness, which, in the opinion of the Investigators would compromise participation in the study (e.g. impaired mental capacity, alcoholism
* Any condition which the Investigators judge to preclude safe participation in the study or to confound the evaluation of the study outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
The proportion of participants achieving ≥80% HU adherence as assessed through medication possession ratio. | At the end of 3 months of Hydroxyurea treatment and monitoring.
  The proportion of participants achieving ≥80% HU adherence will compared between the two arms.

SECONDARY OUTCOMES:
Efficacy of Hydroxyurea treatment as measured through the mean change in fetal hemoglobin (%), | At the end of 3 months of Hydroxyurea treatment and monitoring.
  The mean change in fetal hemoglobin (between baseline and end of 3 months) will be compared between the two arms.
The proportion of participants experiencing serious adverse events (SAE) related to hydroxyurea | at week 2, 6 ,10 and at the end of 3 months of Hydroxyurea treatment and monitoring.
  The overall proportion of participants experiencing SAE during the 3 months of Hydroxyurea treatment will be evaluated as a measure of the safety of treatment with Hydroxyurea

OTHER OUTCOMES:
Incidence of laboratory adverse events, fever and other sickle cell anemia symptoms | At the end of 3 months Hydroxyurea treatment and monitoring
  The incidence during 3 months of treatment will be compared with the incidence during pre-treatment period
Level of leucopenia in relation to incidence rates of fever as indicator of possible infection | At the end of 3 months Hydroxyurea treatment and monitoring
  The level of leucopenia in relation to incidence rate of fever during 3 months of treatment with be compared with that during the pre-treatment period
Mean change in estimated glomerular filtration rate as a measure of kidney function | At the end of 3 months Hydroxyurea treatment and monitoring
  The mean change in estimated glomerular filtration rate will be evaluated as an indicator of deteriorating renal function after Hydroxyurea exposure
Mean change in the level of Lactate Dehydrogenase (LDH) from baseline | At the end of 3 months Hydroxyurea treatment and monitoring
  Serum LDH level (U/L) is usually elevated in sickle cell anemia indicating hemolysis. A decrease in the level of LDH will be considered favorable effect of Hydroxyurea
Mean change in reticulocyte count from baseline | At the end of 3 months Hydroxyurea treatment and monitoring
  Reticulocyte count is usually increased in sickle cell anemia, indicating of hemolysis (a decrease in reticulocyte count % will be considered favorable effect of Hydroxyurea)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Makani, PhD, Study Chair — Muhimbili University of Health and Allied Sciences; Abel Makubi, MMed, Principal Investigator — Muhimbili University of Health and Allied Sciences; Philip Sasi, PhD, Study Director — Muhimbili University of Health and Allied Sciences
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Yes, investigators plan to share the database with one of the collaborators, University of Pittsburgh, USA

REFERENCES:
- [Derived] Makubi A, Sasi P, Ngaeje M, Novelli EM, Mmbando BP, Gladwin MT, Makani J. Rationale and design of mDOT-HuA study: a randomized trial to assess the effect of mobile-directly observed therapy on adherence to hydroxyurea in adults with sickle cell anemia in Tanzania. BMC Med Res Methodol. 2016 Oct 18;16(1):140. doi: 10.1186/s12874-016-0245-9. PMID 27756209